CLINICAL TRIAL: NCT01670435
Title: Assessment of the Safety and Efficacy of Ciproxan-I.V. in Daily Clinical Practice - Analysis Results From a Post-marketing Surveillance
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Medical Director, Bayer Yakuhin, Ltd.
Other Study IDs: 15029; CIPRO-IV-2007 (Other: company internal)
Record Dates: First submitted 2012-08-07; First posted 2012-08-22 (Estimated); Last update posted 2012-08-28 (Estimated); Status verified 2012-08

CONDITIONS: Infection
Keywords: Ciprofloxacin; sepsis; infection; pneumonia; peritonitis; cholecystitis; cholangitis; anthrax
MeSH Terms: conditions — Infections; Sepsis; Pneumonia; Peritonitis; Cholecystitis; Cholangitis; Anthrax | interventions — Ciprofloxacin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Ciprofloxacin (BAYQ3939)

INTERVENTIONS:
Drug: Ciprofloxacin (BAYQ3939) — Patient treated with Ciproxan as a first line treatment in daily clinical practice

SUMMARY:
This study is a post-marketing surveillance in Japan, and it is a local prospective and observational study of patients who have received Ciproxan intravenously as a first-line treatment for sepsis, secondary skin infections followed by superficial burn, post-surgical or post-traumatic, pneumonia, peritonitis, cholecystitis, cholangitis, anthrax. The objective of this study is to assess safety and efficacy of Ciproxan in daily clinical practice. A total of 3,000 patients are to be enrolled and assessed during the period of treatment with Ciproxan.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received Ciproxan as a first-line treatment were eligible for the study, among those with sepsis, secondary infection due to trauma, burn, or surgical wound, pneumonia, peritonitis, cholecystitis, cholangitis, and anthrax as the indications of this drug.

Exclusion Criteria:

* Patients who are contraindicated based on the product label.

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who received Ciproxan as a first-line treatment were eligible for the study, among those with sepsis, secondary infection due to trauma, burn, or surgical wound, pneumonia, peritonitis, cholecystitis, cholangitis, and anthrax as the indications of this drug.
Sampling Method: Non-Probability Sample
Enrollment: 3274 (Actual)
Dates: Start 2007-05; Primary Completion 2010-06 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse drug reactions (ADRs) and serious adverse events (AEs) | After 9 days
Clinical efficacy by four grade (Response, Minor Response, No Response, and Indeterminable) at an investigator discretion | After 9 days

SECONDARY OUTCOMES:
ADR incidence rates classified by patient's background factors | After 9 days
Efficacy rate calculated with Response and Minor Response considered as responder | After 9 days
Efficacy rates classified by patient's background factors | After 9 days

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Japan